CLINICAL TRIAL: NCT00179920
Title: Chemotherapy Plus Local Surgical Treatment in Children With Intraocular Germ-Line Retinoblastoma
Brief Title: Chemotherapy Treatment for Children With Intraocular Germ-Line Retinoblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Stewart Goldman, Division Head, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS 0294
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Retinoblastoma; Retinal Neoplasms
MeSH Terms: conditions — Retinoblastoma; Retinal Neoplasms | interventions — Carboplatin; Etoposide; Cryotherapy

INTERVENTIONS:
Drug: Carboplatin
Drug: VP-16
Procedure: Local Surgery
Procedure: Cryotherapy
Procedure: Laser hyperthermia

SUMMARY:
Retinoblastoma is an unusual cancer of early childhood involving tumor is both eyes or, in certain circumstances, one eye only. This condition is the result of an abnormal gene which makes both retinas (the back of the eye) vulnerable to develop multiple tumors. Growths in the eye impair vision temporarily or permanently. These tumors are malignant, which means that they can grow within the eye, spread outside of the eye, and be fatal if untreated.

Standard therapy for bilateral retinoblastoma includes removal of one eye if vision cannot be save and radiation treatment of either eye in which vision might be saved. Radiation controls tumor growth in the majority of cases. Another standard method is cryotherapy (freezing a tumor to kill it). Chemotherapy (medicines used to kill tumor cells) has been used in the past for tumor in or outside the eye, but is not standard. Hyperthermia, increasing the temperature of a tumor to kill it, is widely performed, and can be done to a retinoblastoma tumor by a laser; this method is not standard.

The problem with removal of an eye is that any hope of vision is lost. The problems with radiation include incomplete control of tumor, injury to the eye or surrounding tissue with decreased growth, and that (due to the abnormal retinoblastoma gene) children are very susceptible to develop other tumors, especially in the tissue which was given radiation.

The doctors at Children's Memorial Hospital are using a newer form of treatment, including laser hyperthermia, chemotherapy and cryotherapy to decrease retinoblastoma tumors. Some may be controlled indefinitely, reducing the number of eyes that need radiation or removal.

OBJECTIVES

1. To find out how well chemotherapy plus cryotherapy and laser hyperthermia work on retinoblastoma tumors.
2. To find out whether vision can be saved and tumors controlled without radiation or removal of the eye.

ELIGIBILITY:
Eligibility Criteria:

* Initial clinical diagnosis of Retinoblastoma, with Bilateral tumors, OR Unilateral tumor with hope for salvage of vision AND Multiple primary tumors, or positive family history for retinoblastoma, or age < 12 months
* No prior antitumor therapy (except enucleation of one eye)
* At least one tumor exceeds 6 mm in diameter
* No evidence of dissemination outside the globe
* Signed IRB-approved informed consent
* Patient/family available for follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1996-04; Study Completion 2006-09

PRIMARY OUTCOMES:
To determine if a multimodal approach can provide durable control of retinoblastoma and specifically:
Estimate the proportion of eyes in which radiation therapy can be omitted
Estimate the proportion of eyes in which vision can be retained

SECONDARY OUTCOMES:
To estimate the response rate and duration for primary retinoblastoma tumors to combination therapy with carboplatin and VP-16
To estimate the response rate of qualifying in situ retinoblastoma tumors to local surgical therapies, specifically estimate tumor response and duration after laser hyperthermia concurrent with carboplatin
Estimate tumor response and duration after cryotherapy
To estimate the control rate of vitreous involvement by retinoblastoma to carboplatin and VP-16
To detect any toxicities resulting from multimodal therapy plus local surgical options

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Goldman, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States